CLINICAL TRIAL: NCT01570439
Title: To Identify HLA-A1101-restricted Peptide Epitopes Derived From Novel Oncoantigens (URLC10, KIF20A, and CDCA1) Applicable for Cancer Vaccine in Singapore
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: KK001
Record Dates: First submitted 2012-04-02; First posted 2012-04-04 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Anonymous Donors at Blood Donation Center (NUH)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Aim: To identify HLA-A1101-restricted peptide epitopes derived from novel Oncoantigens (URLC10, KIF20A, and CDCA1) applicable for Cancer Vaccine in Singapore.

Methods: The panel of candidate peptides are synthesized and tested for their ability to induce peptide-specific CTL responses, in order to screen the peptide epitopes applicable for the cancer vaccination. Briefly, peripheral blood lymphocytes (PBLs) derived from HLA-A1101(+) healthy donors are taken and cultured in the presence of the each candidate peptide with recombinant IL-2 for 2 weeks, and then, re-stimulated with dendritic cell pulsed with the peptide following another 2 week culture. Thereafter, CD8(+) T lymphocytes were negatively selected with CD4-magnetic beads from cultured lymphocytes and tested for their peptide specificity employing enzyme-linked immunospot (ELISPOT) assay. These conditions are completely performed in in-vitro system. Importance in medicine: If one could identify the peptide epitopes from novel Oncoantigens, it is applicable for clinical trials of cancer vaccination.

Benefits & Risks : There is no risk except for the matter of venipuncture in each individuals.

The ideal target molecules for cancer vaccination are thought to be selectively expressed in tumor cells, but not in the normal cells, with high frequent and homogenous expression within tumor. We have proved that novel Oncoantigens, URLC10, KIF20A and CDCA1, have these characters as ideal target molecules for the cancer vaccination and are highly expressed in a variety of tumor type such as gastric, lung, and pancreas cancer. Since HLA-A1101 haplotype is most frequent in Singaporean, it is essential to indentify the HLA-A1101-restriced peptides derived from these Oncoantigens to develop cancer vaccination.

ELIGIBILITY:
Inclusion Criteria:

* The participants should be healthy,
* non-pregnant adults who weigh at least 50kgs

Exclusion Criteria:

* Age of < 22 and > 80 years old.
* Pregnancy (women of childbearing potential: Refusal or inability to use effective means of contraception)
* Decision of unsuitableness by Principal Investigator or physician-in-charge.

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Anonymous donors at blood donation center in NUH.
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
To identify HLA-A1101-restricted peptide epitopes derived from novel Oncoantigens (URLC10, KIF20A, and CDCA1) applicable for Cancer Vaccine in Singapore.

CONTACTS AND LOCATIONS:
Locations (1):
- Nationa University Hospital, Singapore, Singapore

REFERENCES:
- [Background] Kono K, Mizukami Y, Daigo Y, Takano A, Masuda K, Yoshida K, Tsunoda T, Kawaguchi Y, Nakamura Y, Fujii H. Vaccination with multiple peptides derived from novel cancer-testis antigens can induce specific T-cell responses and clinical responses in advanced esophageal cancer. Cancer Sci. 2009 Aug;100(8):1502-9. doi: 10.1111/j.1349-7006.2009.01200.x. Epub 2009 May 14. PMID 19459850
- [Background] Mizukami Y, Kono K, Daigo Y, Takano A, Tsunoda T, Kawaguchi Y, Nakamura Y, Fujii H. Detection of novel cancer-testis antigen-specific T-cell responses in TIL, regional lymph nodes, and PBL in patients with esophageal squamous cell carcinoma. Cancer Sci. 2008 Jul;99(7):1448-54. doi: 10.1111/j.1349-7006.2008.00844.x. Epub 2008 Apr 30. PMID 18452554